CLINICAL TRIAL: NCT00785421
Title: A Prospective, Randomized Trial Of Simultaneous Pancreatic Cancer Treatment With Enoxaparin and ChemoTherapy (PROSPECT)
Brief Title: Chemotherapy With or Without Enoxaparin in Pancreatic Cancer
Acronym: PROSPECT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CONKO-Studiengruppe (Other)
Collaborators: Sanofi (Industry); Amgen (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Uwe Pelzer MD, Dr. med. Uwe Pelzer, CONKO-Studiengruppe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONKO 004; CCT-NAPN-16752
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Pancreatic Cancer
Keywords: heparin; LMWH; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Enoxaparin; Gemcitabine; Cisplatin; Leucovorin; Fluorouracil; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients with KPS > 80% and normal kidney function receive GFFC + LMWH (gemcitabine 1 g/m2 (30 min), cisplatin 30 mg/m2 (90 min), 5-fluorouracil 750 mg/m2 (24 h), folinic acid 200 mg/m2 (30 min), d1, 8; q3w +/- Enoxaparin 1mg/kg daily s.c.).
  Pts with KPS < 80 % and increased creatinin plasma levels (>1.3 mg/dl) receive the current standard therapy (gemcitabine 1 g/m2 (30 min), d1, 8, 15; q4w) + Enoxaparin 1mg/kg daily s.c.
  After 12 weeks of initial chemotherapy all patients who have not progressed received the standard therapy (gemcitabine mono) + Enoxaparin 40mg/d s.c.
  Interventions: Drug: enoxaparin; Drug: chemotherapy with LMWH - enoxaparin
- B (Active Comparator): Patients with KPS > 80% and normal kidney function receive GFFC - LMWH (gemcitabine 1 g/m2 (30 min), cisplatin 30 mg/m2 (90 min), 5-fluorouracil 750 mg/m2 (24 h), folinic acid 200 mg/m2 (30 min), d1, 8; q3w - Enoxaparin 1mg/kg daily s.c.).
  Pts with KPS < 80 % and increased creatinin plasma levels (>1.3 mg/dl) receive the current standard therapy (gemcitabine 1 g/m2 (30 min), d1, 8, 15; q4w) - Enoxaparin 1mg/kg daily s.c.
  After 12 weeks of initial chemotherapy all patients who have not progressed received the standard therapy (gemcitabine mono) - Enoxaparin 40mg/d s.c.
  Interventions: Drug: only chemotherapy

INTERVENTIONS:
Drug: enoxaparin — Patients receive GFFC +/- LMWH (gemcitabine 1 g/m2 (30 min), cisplatin 30 mg/m2 (90 min), 5-fluorouracil 750 mg/m2 (24 h), folinic acid 200 mg/m2 (30 min), d1, 8; q3w +/- Enoxaparin 1mg/kg daily s.c.). Pts with KPS < 80 % and increased creatinin plasma levels (>1.3 mg/dl) receive the current standard therapy (gemcitabine 1 g/m2 (30 min), d1, 8, 15; q4w) +/- LMWM +/- Enoxaparin 1mg/kg daily s.c. After 12 weeks of initial chemotherapy all patients who have not progressed received the standard therapy (gemcitabine mono) +/- Enoxaparin 40mg/d s.c.
  Other Names: gemcitabine; cisplatin; folinic acid; 5-FU
  Arms: A
Drug: chemotherapy with LMWH - enoxaparin — 1-12 weeks: enoxaparin 1g/m², s.c. 12-PD or event: enoxaparin 0,4g s.c.
  Other Names: gemcitabine; cisplatin; folinic acid; 5-FU
  Arms: A
Drug: only chemotherapy — observation, no treatment with LMWH
  Other Names: gemcitabin; cisplatin; folinic acid; 5-FU
  Arms: B

SUMMARY:
To evaluate the safety and efficacy of chemotherapy with or without enoxaparin. This study is powered to decrease the DVT/ VTE events rate from 10% to 3% with enoxaparin in the experimental arm.

N=540pts, dropout-rate 15%, power 80 %, two sided, significant level 5%

DETAILED DESCRIPTION:
Approximately 20% of patients (pts) diagnosed with pancreatic adenocarcinoma (PA) develop venous thromboembolism, which may contribute to the dismal prognosis of PA. A small phase II trial suggested an improved survival by the addition of low molecular weight heparin (LMWH) to chemotherapy. We conducted a small pilot study which indicated that the addition of enoxaparin to chemotherapy GFFC chemotherapy is safe and feasible in pts with advanced PA. Furthermore, results of several phase III studies suggest that pts in good performance status may benefit from more intensive chemotherapy regimen (Riess et al; Heinemann et al; ASCO 2005). Based on these considerations we started the multicenter phase III study CONKO 004.

540 patients are to be recruited into this study. Primary stratification takes place according to Karnofsky performance status and kidney function. Patients with KPS > 80% and normal kidney function receive GFFC +/- LMWH (gemcitabine 1 g/m2 (30 min), cisplatin 30 mg/m2 (90 min), 5-fluorouracil 750 mg/m2 (24 h), folinic acid 200 mg/m2 (30 min), d1, 8; q3w +/- Enoxaparin 1mg/kg daily s.c.). Pts with KPS < 80 % and increased creatinin plasma levels (>1.3 mg/dl) receive the current standard therapy (gemcitabine 1 g/m2 (30 min), d1, 8, 15; q4w) +/- LMWM +/- Enoxaparin 1mg/kg daily s.c. After 12 weeks of initial chemotherapy all patients who have not progressed received the standard therapy (gemcitabine mono) +/- Enoxaparin 40mg/d s.c.

ELIGIBILITY:
Inclusion Criteria:

* histological or cytological pancreatic carcinoma, stage IV A, b
* no preceding radio or chemotherapy of the primarius or the reference lesions
* Karnofsky performance status ≥ 60%
* measurable tumor lesion by spiral CT or MRT not older than 14 days
* no deep venous thrombosis within the last 2 years
* patient compliance and geographical proximity of the residence, which make an adequate follow up possible
* sufficient bone marrow reserve: leukocyte ≥ 3.5 × 109 /l, thrombocyte ≥ 100 × 109 /l
* signed informed consent
* minimum age of 18 years
* women/men must provide sufficient pregnancy prevention

Exclusion Criteria:

* preexisting indication for anti-coagulation of other reason
* bleeding in the last 2 weeks or increased bleeding risk (e.g. serious coagulating disturbance, active stomach or intestine ulzera, or had operational interferences in the last 2 weeks)
* body weight < 45 kg and/or > 100 kg
* pregnancy or insufficient preventing methods in the study process
* serious illness, which are incompatible with a study participation
* hypersensitivity to study drugs
* patients with serious kidney malfunction (Creatininclearance < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
DVT/TVE event rate | After 12 events and after 24 events or after 540 pts recruited

SECONDARY OUTCOMES:
TTP, OS, side effects | after 12 events and after 24 events or after 540 pts are recruited

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Riess, PHD, Study Director — CONKO Study Group
Locations (1):
- Universitätsmedizin - Berlin - Charite, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539